CLINICAL TRIAL: NCT06337604
Title: A Phase 1, Single-center, Double-blind, Randomized, Placebo-controlled Clinical Trial to Evaluate the Safety and Tolerability, Pharmacokinetics, and Preliminary Efficacy of Multiple Administrations of TNP-2092 Capsules in Combination With Rabeprazole Sodium Enteric-coated Tablets in Asymptomatic Healthy Subjects With Helicobacter Pylori Infection
Brief Title: The Safety and Tolerability, Pharmacokinetics of TNP-2092 Capsules in Combination With Rabeprazole Sodium Enteric-coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2092-04
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — TNP-2092

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Rabeprazole sodium enteric-coated tablets + TNP-2092 capsules (n = 10)
  Interventions: Drug: TNP-2092 capsules; Drug: Rabeprazole sodium enteric-coated tablets
- Control Group (Placebo Comparator): Rabeprazole sodium enteric-coated tablets + TNP-2092 capsules placebo (n = 10)
  Interventions: Drug: TNP-2092 capsules placebo; Drug: Rabeprazole sodium enteric-coated tablets

INTERVENTIONS:
Drug: TNP-2092 capsules — TNP-2092 capsules 300 mg twice daily(BID): Taken with 240 mL of warm water 30 minutes (± 5 minutes) after breakfast and dinner, with a 12-hour interval between the two doses. Such administration will last 14 consecutive days. The last administration will be on the morning of Day 15. There will be a total of 29 doses.
  Other Names: Rifaquizinone
  Arms: Study Group
Drug: TNP-2092 capsules placebo — TNP-2092 Capsules Placebo 300 mg BID : Taken with 240 mL of warm water 30 minutes (± 5 minutes) after breakfast and dinner, with a 12-hour interval between the two doses. Such administration will last 14 consecutive days. The last administration will be on the morning of Day 15. There will be a total of 29 doses.
  Arms: Control Group
Drug: Rabeprazole sodium enteric-coated tablets — Rabeprazole sodium enteric-coated tablets (20 mg BID): Taken with 240 mL of warm water 30 minutes (± 5 minutes) before breakfast and dinner for 14 consecutive days. The last administration will be on the morning of Day 15. There will be a total of 29 doses.

SUMMARY:
A phase 1, single-center, double-blind, randomized, placebo-controlled clinical trial to evaluate the safety and tolerability, pharmacokinetics, and preliminary efficacy of multiple administrations of TNP-2092 Capsules in combination with Rabeprazole Sodium Enteric-coated Tablets in asymptomatic healthy subjects with Helicobacter pylori infection

ELIGIBILITY:
Inclusion Criteria:

* Those who have signed the Informed Consent Form before the trial, and fully understand the trial content, procedures, and possible adverse reactions.
* Those who are able to complete the study according to the requirements of the protocol.
* Subjects (including male subjects) who agree to have no pregnancy plan and voluntarily take effective contraceptive measures from the screening date to 6 months after the last administration of the investigational product.
* Sex: male or female.
* Age: 18 - 50 years (inclusive).
* BMI: 18.0 - 28.0 kg/m2 (inclusive).
* Subjects who do not smoke, or have smoked less than 5 cigarettes per day within 3 months before screening; subjects who do not drink alcohol, or have drunk less than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) within 6 months before screening; subjects who have not smoked or drunk alcohol within 48 hours before admission to the study site.
* Subjects whose clinical laboratory test results are within the normal range or whose test results are abnormal but judged by the investigator to be of no clinical significance.
* Subjects with a positive 14C urea breath test(UBT) result.

Exclusion Criteria:

* Subjects with an allergic constitution, a history of allergic diseases or a history of drug allergy.
* Subjects with a history of alcohol or drug abuse in the past 10 years.
* Subjects who have donated blood within 3 months before enrollment.
* Subjects with regular use of any prescription/over-the-counter drugs, including vitamins, minerals, nutritional supplements or herbs, within 2 weeks before enrollment and during the study period.
* Subjects who have taken any drug that changes the activity of liver enzymes 28 days before taking the investigational product or during the study.
* Subjects who have participated in any clinical trials within 3 months before enrollment.
* Subjects with a history of eradication of Helicobacter pylori.
* Subjects who are suffering or have suffered from digestive tract diseases, including digestive tract ulcer, etc.
* Subjects with symptoms or past medical history of cardiovascular, respiratory, urinary, neurological, blood, immune, endocrine system diseases or tumor, mental illness, or any situation which, in the opinion of the investigator, may threaten the safety of the subjects or affect the correctness of the trial results.
* Subjects whose blood pressure remains above 150/95 mmHg after retest.
* Pregnant or lactating women.
* Subjects who are HIV positive, syphilis positive, hepatitis B surface antigen positive, hepatitis C antibody positive.
* Subjects who have had caffeinated beverages or foods (coffee, tea, coke, chocolate and energy drinks), grapefruit (fruit juice) and alcohol within 48 hours (2 days) before the clinical study.
* Other circumstances deemed by the investigator to be unsuitable for the subject to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) | Within 15 minutes before the morning dose of Rabeprazole Sodium Enteric-coated Tablets, and 20 minutes, 50 minutes, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 8, 10 and 12 hours after the morning dose of Rabeprazole Sodium Enteric-coated Tablets
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods
Area Under the Plasma Concentration Versus Time Curve from 0 to the Last Measurable Concentration (AUC0-t) | Within 15 minutes before the morning dose of Rabeprazole Sodium Enteric-coated Tablets, and 20 minutes, 50 minutes, 1.5, 2.5, 3.5, 4.5, 5.5, 6.5, 8, 10 and 12 hours after the morning dose of Rabeprazole Sodium Enteric-coated Tablets
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Maximum Observed Plasma Concentration (Cmax) of TNP-2092 | Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after administration]
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay at specified time points
Percentage of Participants With Adverse Events (AEs) | Day 1 to Day 49
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China